CLINICAL TRIAL: NCT01507779
Title: Evaluation of The Safety and Immunogenicity of an Influenza A/H1N1 Vaccine (IVACFLU), Produced by IVAC, in Healthy Adults in Vietnam
Brief Title: Safety Trial of Monovalent Whole Virus Influenza (H1N1) Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Institute of Vaccines and Medical Biologicals, Vietnam (Industry); Pasteur Institute, Ho Chi Minh City (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVAC-mH1N1-01
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Influenza vaccine (Experimental): Received 0.50 mL of inactivated monovalent influenza vaccine (IVACFLU), administered intramuscularly, on days 0 and 21
  Interventions: Biological: IVACFLU
- Placebo (Placebo Comparator): Received placebo, administered intramuscularly, on days 0 and 21
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IVACFLU — IVACFLU is a whole virus vaccine, collected in a linear sucrose density gradient solution using a continuous flow centrifuge Alfpa Wassmann and inactivated with formaldehyde. It was formulated to contain 15 mcg hemagglutinin (HA) of influenza A/California/07/2009(H1N1)-like virus per 0.5 mL dose and filled in single dose vials.
  Other Names: whole virion monovalent A/H1N1 influenza vaccine
  Arms: Influenza vaccine
Other: Placebo — Phosphate buffered saline (PBS), pH 7.2, in 0.5 ml single-dose vials.
  Arms: Placebo

SUMMARY:
The study hypothesis is that two 0.5 ml doses of non-adjuvanted whole virion monovalent A/H1N1 influenza vaccine (IVACFLU)--each dose with an HA content of 15 mcg from A/California/07/2009 (H1N1)-like virus--will be safe and immunogenic in healthy adults.

DETAILED DESCRIPTION:
This is a phase I, double-blind, individually-randomized (1:1, vaccine:placebo), controlled trial with two groups, IVACFLU (A/H1N1) and placebo. Healthy male and female adults 18 through 40 years of age will be invited to participate. In addition to sponsor monitoring of safety, Program for Appropriate Technology in Health (PATH) will review safety data. Safety data through 7 days post-dose one for all subjects will be reviewed in a blinded fashion prior to administration of dose two of study vaccine or placebo. PATH will review all adverse events (AEs), including clinical laboratory evaluations (pre- and post-vaccination) and will advise if the volunteers may receive dose two of study vaccine or placebo. For all subjects, the procedures and timelines are summarized below.

On the day of first screening (S1), about 14 days (between 5 and 30 days) prior to administration of dose one of study vaccine or placebo, subjects will be screened for eligibility through medical history review, physical examination, testing for serologic evidence of chronic viral infection [human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV)], routine biochemical and hematological blood tests and urinalysis by dipstick. For screening for serologic evidence of chronic viral infections, appropriate pre- and post-test counseling must be provided.

Subject screening for eligibility will continue and be completed on the second screening day (S2). This second screening day will occur the same day as scheduled enrollment into the trial and administration of study vaccine or placebo (Day 0). Women will undergo pregnancy tests using urine samples on Day 0. Fully eligible subjects will be enrolled into the trial. At that time, blood specimens will be collected for immunological testing prior to administration of study vaccine or placebo. Subjects will be unaware of which allocation, IVACFLU or placebo, is received; study vaccine and placebo will be masked. Subjects will be carefully monitored for adverse reactions for 60 minutes after vaccination.

During the first week following vaccination, subjects will be asked to record local and general signs and symptoms using preprinted diary cards, thermometer, and small ruler. Concomitant medications will also be recorded. In addition to solicited signs, subjects will be asked to report any other adverse events, whether or not they believe that the event is related to the vaccination. Member of the investigator's clinical team will visit subjects one and five days after vaccination to check that subjects are correctly completing the diary card and to check on the subjects' well-being. Subjects will then return to the study clinic 7 days after dose one. At that time, the investigator will check the subjects' diary cards and transcribe all adverse events onto the case report forms using medical language. Blood and urine specimens will also be collected for routine biochemical and hematological blood tests and urinalysis by dipstick.

Two days before subjects are scheduled to receive dose two, subjects will be visited or called to remind them of the next visit to the study clinic and to check on the subjects' well-being. Subjects will return to the study clinic at 3 weeks after administration of dose one of study vaccine or placebo in order to receive dose two. At that time, interim histories and concomitant medications will be reviewed. Women will again undergo urine pregnancy tests. All subjects will undergo collection of blood and urine specimens for routine biochemical and hematological blood tests and urinalysis by dipstick and collection of blood serum specimens for immunologic analyses. Then subjects will receive dose two of study vaccine or placebo and be monitored for 60 minutes.

After receipt of dose two, subjects will again complete diary cards for 7 days after vaccination with visits by members of the investigator's clinical team again at days one and five after vaccination to check that the subjects are correctly completing diary cards and to check on the subjects' well-being. Subjects will then return to the study clinic 7 days after dose two (Day 28) for review of diary cards by the investigator and collection of blood and urine specimens for routine biochemical and hematological blood tests and urinalysis by dipstick.

Two days before the subjects' next scheduled visit at 3 weeks after administration of dose two, subjects will be visited or called to remind them of the next visit to the study clinic and to check on the subjects' well-being. Subjects will then return to the study clinic at 3 weeks after administration of dose two (Day 42) of study vaccine or placebo for another study visit. At that time, interim histories and concomitant medications will again be reviewed and final blood specimens will be collected for immunogenicity analyses. Women will also undergo a final pregnancy screen.

Subjects will then be asked to immediately report severe adverse events (SAEs) which occur from Day 42 to Day 201 (approximately 6 months after receipt of dose two). To facilitate this reporting, a member of the investigator's team will visit or call the subjects monthly to check on their well-being. At last study visit on Day 201, subjects will be interviewed and examined one last time before completing the study.

For the evaluation of serum antibodies (by hemagglutination inhibition and microneutralization), serum specimens will be collected on Day 0 (prior to administration of dose one of study vaccine or placebo), on Day 21 (prior to administration of dose two of study vaccine or placebo) and on Day 42.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult 18 (age of legal consent in Vietnam) through 40 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* Free of obvious health problems, as established by the medical history and screening evaluations, including physical examination.
* Capable and willing to complete diary cards and willing to return for all follow-up visits
* For females, willing to utilize reliable birth control measures (intrauterine device, birth control pills, condoms) through the Day 42 visit.

Exclusion Criteria:

* Participation in another clinical trial involving any therapy within the previous three months or planned enrollment in such a trial during the period of this study.
* Receipt of any non-study vaccine within four weeks prior to enrollment or refusal to postpone receipt of such vaccines until after the Day 42 visit.
* Current or recent (within two weeks of enrollment) acute illness with or without fever.
* Receipt of immune globulin or other blood products within three months prior to study enrollment or planned receipt of such products prior to the Day 42 visit.
* Chronic administration (defined as more than 14 consecutively-prescribed days) of immunosuppressants or other immune-modulating therapy within six months prior to study enrollment. (For corticosteroids, this means prednisone or equivalent, >=0.5 mg per kg per day; topical steroids are allowed.)
* History of asthma.
* Hypersensitivity after previous administration of any vaccine.
* Other AE following immunization, at least possibly related to previous receipt of any vaccine.
* Suspected or known hypersensitivity to any of the study vaccine components, including chicken or egg protein.
* Known hypersensitivities (allergies) to food or the natural environment.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, metabolic, neurologic, psychiatric or renal functional abnormality, as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives..
* History of leukemia or any other blood or solid organ cancer.
* History of thrombocytopenic purpura or known bleeding disorder.
* History of seizures.
* Known or suspected immunosuppressed or immunodeficient condition of any kind, including HIV infection.
* Known chronic HBV or HCV infection.
* Known active tuberculosis or symptoms of active tuberculosis, regardless of cause.
* History of chronic alcohol abuse and/or illegal drug use.
* Pregnancy or lactation. (A negative pregnancy test will be required before administration of study vaccine or placebo for all women of childbearing potential.)
* History of Guillain-Barre' Syndrome
* Any condition that, in the opinion of the investigator, would increase the health risk to the subject if he/she participates in the study or would interfere with the evaluation of the study objectives.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Neuzil, MD, MPH, Study Director — PATH; Le V Be, MD, PhD, Study Director — Institute of Vaccines and Medical Biologicals, Vietnam; Ho V Thang, MD, MSc, Principal Investigator — Pasteur Institute
Locations (1):
- Ben Luc Health Center, Bến Lức, Long An, Vietnam

REFERENCES:
- [Derived] Thang HV, Huong VM, Victor JC, Van CB, Nga NT, Be LV, Cuong NP, Tsvetnitsky V, Neuzil KM, Power M, Flores J. Safety and immunogenicity of inactivated monovalent influenza A/H1N1 vaccine candidate manufactured in Vietnam. Vaccine. 2018 Nov 12;36(46):6918-6925. doi: 10.1016/j.vaccine.2018.10.013. Epub 2018 Oct 15. PMID 30337172

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Influenza Vaccine | Placebo
Started | 23 | 25
Completed | 23 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Influenza Vaccine | Placebo | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (6.31) | 31.3 (5.11) | 29.9 (5.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 10 | 7 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Kinh | 23 | 25 | 48
Region of Enrollment [Number; unit: participants]
  Vietnam | 23 | 25 | 48
Handedness [Count of Participants; unit: Participants]
  Left-handed | 5 | 2 | 7
  Right-handed | 18 | 23 | 41
Height [Mean (Standard Deviation); unit: centimeters] | 160.5 (6.01) | 156.9 (5.90) | 158.7 (6.16)
Weight [Mean (Standard Deviation); unit: kilograms] | 55.7 (7.76) | 55.1 (7.74) | 55.4 (7.67)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Maximum Systemic Reaction After Vaccination 1
Description: Systemic and local reactogenicity data were collected on Study Days 0, 7, 21 and 28, prevaccination, and within 60 minutes post-vaccination by clinic staff. Subjects completed diary cards for 7 days after each vaccination and received visits from the investigator's clinical team at Days 1 and 5 following each vaccination. Solicited systemic reactogenicity events included body temperature, feverishness, chills, cough, difficulty breathing, runny nose, nasal congestion, sore throat, hoarseness of voice, headache, confusion, convulsions/seizures, fatigue/malaise, muscle aches, joint pain, pink or red eyes, sore eyes, itchy eyes, drainage from eyes, ear pain or discharge, rash, abdominal pain, diarrhea, vomiting and jaundice. Solicited local reactogenicity included size of redness, size of swelling, size of induration, pain, and tenderness.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Influenza Vaccine
Number analyzed (Participants) | 25 | 23
Participants
  Any systemic symptoms: None | 16 | 15
  Any systemic symptoms: Mild | 9 | 6
  Any systemic symptoms: Moderate | 0 | 2
  Feverishness/subjective fever: None | 25 | 22
  Feverishness/subjective fever: Mild | 0 | 1
  Feverishness/subjective fever: Moderate | 0 | 0
  Chills: None | 25 | 23
  Chills: Mild | 0 | 0
  Chills: Moderate | 0 | 0
  Cough: None | 24 | 22
  Cough: Mild | 1 | 1
  Cough: Moderate | 0 | 0
  Difficulty breathing: None | 25 | 22
  Difficulty breathing: Mild | 0 | 1
  Difficulty breathing: Moderate | 0 | 0
  Runny nose: None | 23 | 23
  Runny nose: Mild | 2 | 0
  Runny nose: Moderate | 0 | 0
  Nasal congestion: None | 25 | 23
  Nasal congestion: Mild | 0 | 0
  Nasal congestion: Moderate | 0 | 0
  Sore throat: None | 25 | 23
  Sore throat: Mild | 0 | 0
  Sore throat: Moderate | 0 | 0
  Hoarseness of voice: None | 24 | 23
  Hoarseness of voice: Mild | 1 | 0
  Hoarseness of voice: Moderate | 0 | 0
  Headache: None | 22 | 19
  Headache: Mild | 3 | 2
  Headache: Moderate | 0 | 2
  Confusion: None | 25 | 23
  Confusion: Mild | 0 | 0
  Confusion: Moderate | 0 | 0
  Seizure: None | 25 | 23
  Seizure: Mild | 0 | 0
  Seizure: Moderate | 0 | 0
  Fatigue/malaise: None | 23 | 20
  Fatigue/malaise: Mild | 2 | 3
  Fatigue/malaise: Moderate | 0 | 0
  Muscle aches (generalized): None | 24 | 21
  Muscle aches (generalized): Mild | 1 | 2
  Muscle aches (generalized): Moderate | 0 | 0
  Joint pain: None | 25 | 23
  Joint pain: Mild | 0 | 0
  Joint pain: Moderate | 0 | 0
  Pink or red eyes: None | 25 | 23
  Pink or red eyes: Mild | 0 | 0
  Pink or red eyes: Moderate | 0 | 0
  Sore eyes: None | 25 | 22
  Sore eyes: Mild | 0 | 1
  Sore eyes: Moderate | 0 | 0
  Itchy eyes: None | 25 | 23
  Itchy eyes: Mild | 0 | 0
  Itchy eyes: Moderate | 0 | 0
  Drainage from eyes: None | 25 | 23
  Drainage from eyes: Mild | 0 | 0
  Drainage from eyes: Moderate | 0 | 0
  Ear pain or discharge: None | 25 | 23
  Ear pain or discharge: Mild | 0 | 0
  Ear pain or discharge: Moderate | 0 | 0
  Rash: None | 24 | 22
  Rash: Mild | 1 | 1
  Rash: Moderate | 0 | 0
  Abdominal pain: None | 25 | 23
  Abdominal pain: Mild | 0 | 0
  Abdominal pain: Moderate | 0 | 0
  Diarrhea: None | 24 | 22
  Diarrhea: Mild | 1 | 1
  Diarrhea: Moderate | 0 | 0
  Vomiting: None | 25 | 23
  Vomiting: Mild | 0 | 0
  Vomiting: Moderate | 0 | 0
  Jaundice: None | 25 | 23
  Jaundice: Mild | 0 | 0
  Jaundice: Moderate | 0 | 0

2. Primary Outcome: Number of Participants With Maximum Systemic Reaction After Vaccination 2
Description: as for outcome 1
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Influenza Vaccine
Number analyzed (Participants) | 25 | 23
Participants
  Any systemic symptoms: None | 13 | 19
  Any systemic symptoms: Mild | 10 | 3
  Any systemic symptoms: Moderate | 2 | 1
  Feverishness/subjective fever: None | 25 | 21
  Feverishness/subjective fever: Mild | 0 | 1
  Feverishness/subjective fever: Moderate | 0 | 1
  Chills: None | 25 | 23
  Chills: Mild | 0 | 0
  Chills: Moderate | 0 | 0
  Cough: None | 24 | 20
  Cough: Mild | 1 | 3
  Cough: Moderate | 0 | 0
  Difficulty breathing: None | 25 | 23
  Difficulty breathing: Mild | 0 | 0
  Difficulty breathing: Moderate | 0 | 0
  Runny nose: None | 20 | 21
  Runny nose: Mild | 5 | 1
  Runny nose: Moderate | 0 | 1
  Nasal congestion: None | 23 | 22
  Nasal congestion: Mild | 1 | 1
  Nasal congestion: Moderate | 1 | 0
  Sore throat: None | 23 | 23
  Sore throat: Mild | 1 | 0
  Sore throat: Moderate | 1 | 0
  Hoarseness of voice: None | 25 | 23
  Hoarseness of voice: Mild | 0 | 0
  Hoarseness of voice: Moderate | 0 | 0
  Headache: None | 20 | 21
  Headache: Mild | 3 | 1
  Headache: Moderate | 2 | 1
  Confusion: None | 25 | 23
  Confusion: Mild | 0 | 0
  Confusion: Moderate | 0 | 0
  Seizure: None | 25 | 23
  Seizure: Mild | 0 | 0
  Seizure: Moderate | 0 | 0
  Fatigue/malaise: None | 23 | 23
  Fatigue/malaise: Mild | 2 | 0
  Fatigue/malaise: Moderate | 0 | 0
  Muscle aches (generalized): None | 24 | 22
  Muscle aches (generalized): Mild | 1 | 1
  Muscle aches (generalized): Moderate | 0 | 0
  Joint pain: None | 25 | 23
  Joint pain: Mild | 0 | 0
  Joint pain: Moderate | 0 | 0
  Pink or red eyes: None | 25 | 22
  Pink or red eyes: Mild | 0 | 1
  Pink or red eyes: Moderate | 0 | 0
  Sore eyes: None | 24 | 23
  Sore eyes: Mild | 1 | 0
  Sore eyes: Moderate | 0 | 0
  Itchy eyes: None | 25 | 22
  Itchy eyes: Mild | 0 | 1
  Itchy eyes: Moderate | 0 | 0
  Drainage from eyes: None | 25 | 23
  Drainage from eyes: Mild | 0 | 0
  Drainage from eyes: Moderate | 0 | 0
  Ear pain or discharge: None | 25 | 23
  Ear pain or discharge: Mild | 0 | 0
  Ear pain or discharge: Moderate | 0 | 0
  Rash: None | 22 | 22
  Rash: Mild | 3 | 1
  Rash: Moderate | 0 | 0
  Abdominal pain: None | 25 | 23
  Abdominal pain: Mild | 0 | 0
  Abdominal pain: Moderate | 0 | 0
  Diarrhea: None | 25 | 23
  Diarrhea: Mild | 0 | 0
  Diarrhea: Moderate | 0 | 0
  Vomiting: None | 25 | 23
  Vomiting: Mild | 0 | 0
  Vomiting: Moderate | 0 | 0
  Jaundice: None | 25 | 23
  Jaundice: Mild | 0 | 0
  Jaundice: Moderate | 0 | 0

3. Primary Outcome: Number of Participants With Maximum Local Reaction After Vaccination 1
Description: Systemic and local reactogenicity data were collected on Study Days 0, 7, 21 and 28, prevaccination, and within 60 minutes post-vaccination by clinic staff. Subjects completed diary cards for 7 days after each vaccination and received visits from the investigator's clinical team at Days 1 and 5 following each vaccination. Solicited local reactogenicity included size of redness, size of swelling, size of induration, pain, and tenderness.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Influenza Vaccine
Number analyzed (Participants) | 25 | 23
Participants
  Any local symptoms: None | 20 | 19
  Any local symptoms: Mild | 5 | 4
  Swollen after injection: None | 24 | 23
  Swollen after injection: Mild | 1 | 0
  Red after injection: None | 24 | 23
  Red after injection: Mild | 1 | 0
  Hardness after injection: None | 24 | 23
  Hardness after injection: Mild | 1 | 0
  Painful feeling after injection: None | 25 | 20
  Painful feeling after injection: Mild | 0 | 3
  Pain when touching to the injection: None | 20 | 21
  Pain when touching to the injection: Mild | 5 | 2

4. Primary Outcome: Number of Participants With Maximum Local Reaction After Vaccination 2
Description: as for outcome 3
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Influenza Vaccine
Number analyzed (Participants) | 25 | 23
Participants
  Any local symptoms: None | 21 | 21
  Any local symptoms: Mild | 4 | 2
  Swollen after injection: None | 25 | 23
  Swollen after injection: Mild | 0 | 0
  Red after injection: None | 24 | 22
  Red after injection: Mild | 1 | 1
  Hardness after injection: None | 25 | 23
  Hardness after injection: Mild | 0 | 0
  Painful feeling after injection: None | 25 | 22
  Painful feeling after injection: Mild | 0 | 1
  Pain when touching to the injection: None | 22 | 23
  Pain when touching to the injection: Mild | 3 | 0

5. Primary Outcome: Unsolicited, Non-serious Adverse Events
Description: Subjects completed diary cards for 7 days after each vaccination and received visits from the investigator's clinical team at Days 1 and 5 following each vaccination. Adverse events were collected throughout the study period, and were graded for severity; however unsolicited adverse events were assessed only for relationship to vaccine if the events were immediate reactions or considered to be serious adverse events.
Time Frame: 7 days after each dose (Day 7 and Day 28)
Measure: Number; unit: adverse events
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 23 | 25
adverse events
  Mild | 5 | 14
  Moderate | 12 | 11

6. Secondary Outcome: Geometric Mean Titer of Hemagglutination-inhibition Antibodies (HAI)
Description: Day 0, 21 and 42 blood samples from study subjects (n=48) were tested. The assay is performed in duplicate wells of 2-fold serial dilutions of serum. The hemagglutination titer was reported as the reciprocal of the highest dilution that caused hemagglutination and was expressed in HA units (HAU)/50μL, calculated as the average of results of duplicate wells.
Time Frame: Day 0, Day 21 and Day 42
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 23 | 25
titer
  Day 0 | 13.5 [8.5 to 21.6] | 11.5 [7.7 to 17.2]
  Day 21 | 306.6 [165.1 to 569.6] | 11.2 [7.7 to 16.3]
  Day 42 | 283.7 [161.7 to 497.5] | 11.8 [8.1 to 17.3]

7. Secondary Outcome: Ratio of Geometric Mean Titer of Hemagglutination-inhibition Antibodies (HAI)
Description: as for outcome 6
Time Frame: Day 0, Day 21 and Day 42
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 23 | 25
ratio
  Day 21/Day 0 | 22.69 [11.0 to 46.64] | 0.97 [0.9 to 1.08]
  Day 42/Day 0 | 20.99 [10.6 to 41.45] | 1.03 [0.8 to 1.17]
  Day 42/Day 21 | 0.93 [0.7 to 1.18] | 1.06 [1.0 to 1.14]

8. Secondary Outcome: Number and Percentage of All Subjects Achieving a Four-fold Rise in Hemagglutination-inhibition Antibodies (HAI)
Description: Day 21 and 42 blood samples from study subjects (n=48) were tested. The assay is performed in duplicate wells of 2-fold serial dilutions of serum. The hemagglutination titer was reported as the reciprocal of the highest dilution that caused hemagglutination and was expressed in HA units (HAU)/50μL, calculated as the average of results of duplicate wells.
Time Frame: Day 21 and Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 23 | 25
Participants
  Day 21: 4-fold rise or higher | 20 | 0
  Day 21: Less than 4-fold rise | 3 | 25
  Day 42: 4-fold rise or higher | 21 | 0
  Day 42: Less than 4-fold rise | 2 | 25
  Day 21 or 42: 4-fold rise or higher | 22 | 0
  Day 21 or 42: Less than 4-fold rise | 1 | 25

9. Secondary Outcome: Number and Percentage of Subjects Achieving a Four-fold Rise in Hemagglutination-inhibition Antibodies (HAI) Among Subjects With Baseline Titer Less Than 40
Description: Day 21 and Day 42 blood samples from study subjects (n=48) were tested. The assay is performed in duplicate wells of 2-fold serial dilutions of serum. The hemagglutination titer was reported as the reciprocal of the highest dilution that caused hemagglutination and was expressed in HA units (HAU)/50μL, calculated as the average of results of duplicate wells.
Time Frame: Day 21 and Day 42
Population: Subjects with baseline titer <40
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 17 | 18
Participants
  Day 21: 4-fold rise or higher | 15 | 0
  Day 21: Less than 4-fold rise | 2 | 18
  Day 42: 4-fold rise or higher | 17 | 0
  Day 42: Less than 4-fold rise | 0 | 18

10. Secondary Outcome: Number and Percentage of Subjects Achieving a Four-fold Rise in Hemagglutination-inhibition Antibodies (HAI) Among Subjects With Baseline Titer Greater Than 40
Description: as for outcome 8
Time Frame: Day 21 and Day 42
Population: Subjects with baseline titer >=40
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 6 | 7
Participants
  Day 21: 4-fold rise or higher | 5 | 0
  Day 21: Less than 4-fold rise | 1 | 7
  Day 42: 4-fold rise or higher | 4 | 0
  Day 42: Less than 4-fold rise | 2 | 7

11. Secondary Outcome: Number and Percentage of Subjects Developing a Seroprotective Hemagglutination-inhibition (HAI) Antibody Titer
Description: Seroprotection defined as an HAI titer ≥1:40. Day 21 and 42 blood samples from study subjects (n=48) were tested. The assay is performed in duplicate wells of 2-fold serial dilutions of serum. The hemagglutination titer was reported as the reciprocal of the highest dilution that caused hemagglutination and was expressed in HA units (HAU)/50μL, calculated as the average of results of duplicate wells.
Time Frame: Day 21 and Day 42
Population: Includes subjects who had a baseline titer of <1:40.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 17 | 18
Participants
  Day 21: Response | 15 | 0
  Day 21: No response | 2 | 18
  Day 42: Response | 17 | 1
  Day 42: No response | 0 | 17

12. Secondary Outcome: Geometric Mean Titer of Microneutralizing (MN) Antibodies
Description: Day 0, 21 and 42 specimens were tested in the microneutralization (MN) assay. The microneutralization assay determines the titer of neutralizing antibodies against influenza A/H1N1. The assay is performed in duplicate wells of 2-fold serial dilutions of serum. The 50% neutralizing antibody titer is the reciprocal of the corresponding serum dilution. The geometric mean titers (GMT) and corresponding confidence intervals were based on a log 10 scale.
Time Frame: Day 0, Day 21 and Day 42
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 23 | 25
titer
  Day 0 | 21.2 [11.8 to 38.4] | 17.7 [9.8 to 31.9]
  Day 21 | 595.1 [287.8 to 1230.5] | 18.9 [10.6 to 33.9]
  Day 42 | 725.7 [411.3 to 1280.3] | 18.9 [10.3 to 34.9]

13. Secondary Outcome: Ratio of Geometric Mean Titer of Microneutralization (MN) Antibodies
Description: as for outcome 12
Time Frame: Day 0, Day 21 and Day 42
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 23 | 25
ratio
  Day 21/Day 0 | 28.01 [12.0 to 65.24] | 1.07 [1.0 to 1.20]
  Day 42/Day 0 | 34.16 [16.8 to 69.40] | 1.07 [1.0 to 1.16]
  Day 42/Day 21 | 1.22 [0.9 to 1.61] | 1.00 [0.9 to 1.12]

14. Secondary Outcome: Number and Percentage of All Subjects Achieving a Four-fold Rise in Microneutralization (MN) Antibodies
Description: Day 21 and 42 specimens were tested in the microneutralization (MN) assay. The microneutralization assay determines the titer of neutralizing antibodies against influenza A/H1N1. The assay is performed in duplicate wells of 2-fold serial dilutions of serum. The 50% neutralizing antibody titer is the reciprocal of the corresponding serum dilution. The geometric mean titers (GMT) and corresponding confidence intervals were based on a log 10 scale.
Time Frame: Day 21 and Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 23 | 25
Participants
  Day 21: 4-fold rise or higher | 19 | 0
  Day 21: Less than 4-fold rise | 4 | 25
  Day 42: 4-fold rise or higher | 22 | 0
  Day 42: Less than 4-fold rise | 1 | 25
  Day 21 or 42: 4-fold rise or higher | 22 | 0
  Day 21 or 42: Less than 4-fold rise | 1 | 25

15. Secondary Outcome: Number and Percentage of Subjects Achieving a Four-fold Rise in Microneutralizing (MN) Antibodies Among Subjects With Baseline Titer Less Than 40
Description: as for outcome 8
Time Frame: Day 21 and Day 42
Population: Subjects with baseline titer <40
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 11 | 15
Participants
  Day 21: 4-fold rise or higher | 10 | 0
  Day 21: Less than 4-fold rise | 1 | 15
  Day 42: 4-fold rise or higher | 11 | 0
  Day 42: Less than 4-fold rise | 0 | 15

16. Secondary Outcome: Number and Percentage of Subjects Achieving a Four-fold Rise in Microneutralizing (MN) Antibodies Among Subjects With Baseline Titer Greater Than 40
Description: as for outcome 14
Time Frame: Day 21 and Day 42
Population: Subjects with baseline titer >=40
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 12 | 10
Participants
  Day 21: 4-fold rise or higher | 9 | 0
  Day 21: Less than 4-fold rise | 3 | 10
  Day 42: 4-fold rise or higher | 11 | 0
  Day 42: Less than 4-fold rise | 1 | 10

17. Secondary Outcome: Number and Percentage of Subjects Developing a Seroprotective Microneutralizing (MN) Antibody Titer
Description: Seroprotection defined as an antibody titer of 1:40 or greater. Day 21 and 42 specimens were tested in the microneutralization (MN) assay. The microneutralization assay determines the titer of neutralizing antibodies against influenza A/H1N1. The assay is performed in duplicate wells of 2-fold serial dilutions of serum. The 50% neutralizing antibody titer is the reciprocal of the corresponding serum dilution. The geometric mean titers (GMT) and corresponding confidence intervals were based on a log 10 scale.
Time Frame: Day 21 and Day 42
Population: Includes subjects who had a baseline titer of <1:40.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza Vaccine | Placebo
Number analyzed (Participants) | 11 | 15
Participants
  Day 21: Seroprotection | 9 | 0
  Day 21: No seroprotection | 2 | 15
  Day 42: Seroprotection | 11 | 0
  Day 42: No seroprotection | 0 | 15

ADVERSE EVENTS:
Time Frame: 7 days after each vaccination for non-serious adverse events; 201 days for serious adverse events.
Description: Subjects completed diary cards for 7 days after each vaccination and received visits from the investigator's clinical team at Days 1 and 5 following each vaccination. Additionally, the participant recorded any serious adverse events over the entire study on clinic visits on day 42 and 201.
Arm/Group | Influenza Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 1/25
Other Adverse Events (participants affected / at risk) | 11/23 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine (N=23) | Placebo (N=25)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza Vaccine (N=23) | Placebo (N=25)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 2
Generalized erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Myelopathy (Nervous system disorders) | 0 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 0
Piloerection (Skin and subcutaneous tissue disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rhinitis allergic (Immune system disorders) | 0 | 1
Sciatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No